CLINICAL TRIAL: NCT07040514
Title: 24GUT540: Opportunity for Breast Cancer Patients to Meet With a Pathologist to Review the Pathology Slides of Their Breast Samples
Brief Title: 24GUT540 : Meeting of Breast Cancer Patients and Pathologists
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Edward.J.Gutmann, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Study02002540
Record Dates: First submitted 2025-05-12; First posted 2025-06-27 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: To determine whether meeting with a pathologist to review and discuss the pathologic findings in their breast samples is beneficial to breast cancer patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assessment of Patient understanding of Pathologist input (Other): Assessment of patient understanding of, and sense of control regarding, their disease, and their perception of the potential benefit of having pathologists on their medical team.
  Interventions: Other: Questionnaires of Patient understanding of Pathologist input

INTERVENTIONS:
Other: Questionnaires of Patient understanding of Pathologist input — * Benefit Self-Rating Total Score (assessing patient's perceptions of anticipated and actual extent to which they benefitted from the meeting with the pathologist)
  * Knowledge Questionnaire Total Score (assessing accuracy of knowledge of their own diagnosis and the diagnostic process in general)
  * State-Trait Anxiety Inventory Form Y (Total Scores for state (current) and trait (general) anxiety)

SUMMARY:
Historically, most pathologists have had little direct contact or communication with patients. In the past two decades, however, there has been a modest movement toward patient-pathologist visits in which pathologists review with patients their pathology slides.

Very few studies of such encounters have been conducted. Most surveyed patients reported that the experience was positive and helpful to them. Our basic goal is to determine if such meetings are useful to patients; a secondary goal is to determine if such encounters are useful to, and practical for, pathologists.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age.
2. Patients must have completed initial diagnosis visit with oncologist or surgeon.
3. Must have pathology slides and reports available for review.
4. Must be able to speak English.
5. Must be willing to participate in this research and will be provided with an information sheet.
6. Pregnant women are eligible as this research poses no risk of physical harm to the participant.

Exclusion Criteria:

1. Patients <18 years of age.
2. Patients with DCIS are ineligible.
3. Adults who are unable to provide written signature.
4. Patients from vulnerable patient populations, including infants, minors, those unable to provide informed consent, and those incarcerated or imprisoned at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Participant self-rating of understanding of, and empowerment in relation to, their disease, as measured using pre and post-visit knowledge questionnaires, and survey after meeting with a pathologist. | 1-2 weeks
  Determine understanding improvement from pre-meeting questionnaires and after pathologist visit with post-visit questionnaires, as well as knowledge questionnaire for both timepoints.
  Knowledge Questionnaire: Primary Score: Total Score - Total # correct responses on the knowledge questions (12 items total).
  Survey for Patients after Meeting with Pathologist Primary Score: Item 1 Total Score - Responses will be coded on a 0-4 scale where 0=strongly disagree and 4=strongly agree, and the total will be calculated across items 'a' through 'j' of Item 1.

SECONDARY OUTCOMES:
Participant knowledge of their personal disease characteristics | 1-2 weeks
  Determined by participant completing pre-and-post visit Knowledge Questionnaires.
  Knowledge Questionnaire: Primary Score: Total Score - Total # correct responses on the knowledge questions (12 items total).
Participant general knowledge of breast cancer pathology | 1-2 weeks
  Determined by participant completing pre-and-post visit Knowledge Questionnaires.
  Knowledge Questionnaire: Primary Score: Total Score - Total # correct responses on the knowledge questions (12 items total).

OTHER OUTCOMES:
Participant ratings of helpfulness and other features of meeting with a pathologist such as comfort level with the meeting | 1-2 weeks
  Determined by participant completing post-visit survey.
  Survey for Patients after Meeting with Pathologist Primary Score: Item 1 Total Score - Responses will be coded on a 0-4 scale where 0=strongly disagree and 4=strongly agree, and the total will be calculated across items 'a' through 'j' of Item 1.
Participant anxiety self-rating | 1-2 weeks
  Determined by participant completing State Trait Anxiety Inventory (STAI).
  STAI Form Y-1 contains 40 items, each given a self-reported rating of 1-4, with 1: "Not at all", 2: "Somewhat, 3: "Moderately so", and 4: "Very much so".
Pathologist rating of patient benefit from the meeting and other features of the meeting such as degree to which rapport was established. | 1-2 weeks
  Determined by pathologist completing the post-visit survey.
  Survey for Pathologist After Meeting with Patient Primary Score: Total Score on Items 6 and 7 (8 items total) - Responses will be coded on a 0-4 scale where 0=highly dissatisfied and 4=highly satisfied, and the total will be calculated for items 6 and 7.

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Gutmann, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States